CLINICAL TRIAL: NCT06814873
Title: Enhanced Human Sensorimotor Integration Via Self-modulation of the Somatosensory Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keio University (Other)
Responsible Party: Principal Investigator, Junichi Ushiba, Professor, Keio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-128
Record Dates: First submitted 2025-01-29; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Somatosensory Evoked Potentials, and Electroencephalography
MeSH Terms: interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum (Experimental): Participants in the group received real-time feedback of their own electroencephalogram signal
  Interventions: Behavioral: Neurofeedback
- Sham (Sham Comparator): Participants in the group received feedback of electroencephalogram signal previously recorded from other participants.
  Interventions: Behavioral: Sham-feedback

INTERVENTIONS:
Behavioral: Neurofeedback — The participants received visual feedback of the processed result of neural signals acquired online.
  Arms: Verum
Behavioral: Sham-feedback — Previously recorded neural signals are processed and presented to participants as if the signals from them are processed online.
  Arms: Sham

SUMMARY:
The purpose of this study is to examine the functional and structural modification effects on the brain of a non-invasive experimental device applied to the head and forearms of healthy subjects during motor recall training. The experimental device used in this study is the Brain-Machine Interface (hereinafter referred to as BMI), which is under development in the principal investigator's laboratory. The BMI consists of an arithmetic unit that processes the results in real time using a personal computer, a depth ray that displays the results, a transcutaneous electrical stimulator that is driven based on the results of the arithmetic, and an exoskeletal motor assist device that is driven based on the results of the arithmetic.

DETAILED DESCRIPTION:
This study does not fall under the category of 'medical research involving human subjects' or 'clinical research subject to legal regulations' in Japan, and the appointment of a principal investigator (PI) is not required. For the convenience of registry submission, the name of the principal investigator field has been filled with the name of the study representative (a non-physician).

ELIGIBILITY:
Exclusion Criteria:

* History of neurological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Somatosensory evoked potential | From the timing of pre-training evaluation (before the intervention) to the end of evaluation (after the intervention), with the intervention lasting 30 minutes.
  Median nerve stimulation elicits the somatosensory evoked potentials. Their amplitude was calculated.

SECONDARY OUTCOMES:
Touch typing performance | From the timing of pre-training evaluation (before the intervention) to the end of evaluation (after the intervention), with the intervention lasting 30 minutes.
  A touch typing task was employed to test sensorimotor integration performance

CONTACTS AND LOCATIONS:
Locations (1):
- Keio University, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No